CLINICAL TRIAL: NCT04896398
Title: Effect of Extracorporeal Shock Wave Therapy on Carpal Tunnel Syndrome
Brief Title: The Effect of ESWT in Carpal Tunnel Syndrome
Acronym: ESWT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Ahmet Kivanc Menekseoglu, Principal Investigator, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021-1
Record Dates: First submitted 2021-05-13; First posted 2021-05-21 (Actual); Last update posted 2023-03-20 (Actual); Status verified 2023-03

CONDITIONS: Carpal Tunnel Syndrome
Keywords: ESWT
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Intervention Model Description: After the patients are numbered according to the order of application, they will be divided into 2 groups as study and control groups according to randomization made with the computer program (block randomization). A total of 5 sessions of ESWT (1000 shock, 1.6 bar, 5 Hz) will be applied to the study group (1st group) for 2 weeks. Median nerve and tendon shifting exercises will be taught to the patients and they will be asked to do it regularly. Patients in the control group (Group 2) will be asked to perform median nerve and tendon shifting exercises only for the wrist. Patients will be evaluated before treatment and at 4 and 12 weeks after treatment.
Who Masked: Investigator
Masking Description: The evaluation of the patients will be made by an evaluator who has no knowledge of group distribution.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ESWT Group (Experimental): A total of 5 sessions of ESWT (1000 shock, 1.6 bar, 5 Hz) will be applied to the patients in this group for 2 weeks. Median nerve and tendon shifting exercises will be taught to the patients and they will be asked to do it regularly.
  Interventions: Device: ESWT
- Control Group (No Intervention): Patients in the control group will be asked to do median nerve and tendon shifting exercises only for the wrist.

INTERVENTIONS:
Device: ESWT — In the study group, a total of 5 sessions of focused ESWT (1000 shock, 1.6 bar, 5 Hz) will be applied to the affected wrist within 2 weeks.
  Arms: ESWT Group

SUMMARY:
50 patients who meet the inclusion criteria will be included in this prospective, randomized and controlled study. Demographic information of the patients will be taken and recorded. After the patients are numbered according to the order of application, they will be divided into 2 groups as study and control groups according to randomization with the computer program. A total of 5 sessions of ESWT (1000 shock, 1.6 bar, 5 Hz) will be applied to the study group (1st group) for 2 weeks. Patients will be taught median nerve and tendon shifting exercises and will be asked to do it regularly. Patients in the control group (Group 2) will be asked to perform median nerve and tendon shifting exercises only for the wrist. Patients will be evaluated before treatment, at 4 and 12 weeks after treatment. In the evaluation, Boston Carpal Tunnel Inquiry Form, pain severity assessment with VAS (visual analog scale), neuropathic pain intensity with LANSS scale and median nerve conduction velocity with EMG will be evaluated.

DETAILED DESCRIPTION:
Carpal tunnel syndrome is a clinical picture that occurs with a group of symptoms and signs as a result of compression and compression in the carpal tunnel where the median nerve passes to the wrist. Another name is hand-wrist canal disease, the most common entrapment is neuropathy. It is generally observed in individuals between the ages of 40-60, its prevalence is 4-5%, and it is 3 times more common in women than men. Clinical signs 1.-2.-3. numbness, tingling, abduction and positioning of the thumb, pain in the wrist and inner part of the hand, autonomic symptoms (heat or discoloration, dry skin) worsening of symptoms due to provocative factors (forcing the wrist to flex). Loss of strength and atrophy of the palm muscles occur in the later stages. The diagnosis is made by clinical examination, electrophysiological methods (EMG) and imaging methods (such as ultrasound, magnetic resonance imaging). Clinical examination consists of sensory motor examination and provocative tests. Treatment is divided into conservative and surgical. Among the conservative treatment methods, splinting, exercise (sliding movements of the median nerve and wrist flexor tendons in the wrist), local corticosteroid injection (corticosteroid injection into the carpal tunnel), ultrasound (warming the deep tissues with sound energy), TENS (electrodes placed on the skin). pain relief by applying controlled low-voltage electric current to the nervous system through the skin), paraffin bath (immersion of the hand in a pool of heat-melted paraffin), ergonomic arrangements. ESWT is a widely used treatment method in the treatment of carpal tunnel syndrome in recent years. ESWT is called "Extracorporeal Shock Wave Therapy", in Turkish "Shock Wave Therapy Applied Outside the Body" or simply "Shock Wave Therapy". It is a treatment method based on the principle of focusing the shock (pressure) waves created outside the body to the desired area of the body by means of a steel-headed applicator. Shock waves are single pulsatile acoustic waves of high amplitude. It reaches high pressure (100Mpa) and then negative pressure (5-10 Mpa) in a short time expressed in nanoseconds (10 ns). This device was first applied in the destruction of urinary stones in the 1980s. In the following years, it has been used in cases such as shoulder calcific tendinitis, lateral epicondylitis, plantar fasciitis, and fracture healing. Currently indications for ESWT are non-union fractures, revision arthroplasties, lateral epicondylitis, plantar fascitis, calcified tendinitis of the shoulder, avascular necrosis of the femoral head, Achilles tendinitis, patellar tendinitis, myofascial pain syndrome, ischemic heart disease, peyronia disease, chronic diabetic heart disease. It covers a wide range of disease groups such as ulcers, knee osteoarthritis, complex regional pain syndrome, carpal tunnel syndrome. Studies have shown that ESWT increases angiogenesis, neovascularization, anti-inflammatory growth factor release, progenitor and stem cell activation. Morphological changes were detected in cutaneous sensory nerve fibers with shock wave application on the nerves. It has been observed that there is a relationship between reduction of PGP 9.5 (protein gene product) and CGRP (calcitonin gene-related peptide) and pain reduction following shock application in sensory nerve fibers in the epidermal region. At the same time, integrin molecules are secreted for axonal growth with shock application and this continues cumulatively with ESWT application. GAP 43 (growth associated phosphoprotein) molecule, which is a marker related to axonal regeneration and which is highly expressed especially during neuron development and axonal 3/10 elongation, has been found to increase after ESWT application. In this study, it was aimed to investigate the effectiveness of ESWT treatment applied to patients diagnosed with mild to moderate carpal tunnel syndrome by EMG.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of mild to moderate CTS in the nerve conduction study within the last 1 month,
* Positive Phalen and Tinnel tests in clinical examination
* Who agreed to participate in the study

Exclusion Criteria:

* Patients with cervical radiculopathy,
* Pregnant women,
* Rheumatoid arthritis,
* Thenar atrophy,
* Steroid injection or surgical procedure in the wrist in the last 3 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-11-01 (Actual)

PRIMARY OUTCOMES:
Boston carpal tunnel questionnaire | 3 months
  The functional levels of the patients will be evaluated with the Boston carpal tunnel questionnaire.

SECONDARY OUTCOMES:
Visual Analog Scale | 3 months
  The pain level of the patients will be evaluated with visual analog scale. The visual analog scale is scored between 0 and 10. Increased scores mean more pain.
Median nerve conduction study | 3 months
  Median nerve conduction velocity will be evaluated by ENMG.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmet K Menekşeoğlu, Principal Investigator — Kanuni Sultan Süleyman Research and Training Hospital
Locations (1):
- Ahmet Kıvanç Menekşeoğlu, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Identity information of the patients other than their gender, age and BMI will not be shared.